CLINICAL TRIAL: NCT06450587
Title: Intraocular Pressure Data Collection With Tonometers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icare Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TA032-082
Record Dates: First submitted 2024-05-31; First posted 2024-06-10 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Measurement of IOP Values (Experimental): Measurement of IOP pressure with four different tonometers.
  Interventions: Device: iCare IC1000; Device: iCare ST500; Device: iCare IC200; Device: GAT

INTERVENTIONS:
Device: iCare IC1000 — Measurement of Intraocular Pressure (IOP)
Device: iCare ST500 — Measurement of Intraocular Pressure (IOP)
Device: iCare IC200 — Measurement of Intraocular Pressure (IOP)
Device: GAT — Measurement of Intraocular Pressure (IOP)

SUMMARY:
The goal of this clinical trial is to collect a comprehensive dataset of intraocular pressure values for developing a measurement algorithm for the new hand-held rebound tonometer device. The measurement algorithm shall fulfill the requirements of ANSI Z80.10:2014 standard. The study population is adults (age ≥ 18 years).

The intraocular pressure of the participants will be measured with four different tonometers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Exclusion Criteria:

* Subjects with only one functional eye
* Subjects having poor or eccentric fixation in the study eye(s)
* High corneal astigmatism >3D in the study eye(s)
* Central corneal scarring
* History of prior incisional glaucoma surgery or corneal surgery, including corneal refractive laser surgery in the study eye(s)
* Microphthalmos
* Buphthalmos
* Contact lens use within one week of continuous wear and within one hour if lens is worn occasionally
* Dry eyes (clinically significant)
* Lid squeezers - blepharospasm
* Nystagmus
* Keratoconus
* Any other corneal or conjunctival pathology or infection relevant to this study
* Cataract Extraction within last 2 months in the study eye(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Primary Objective | Through study completion, an average of 4 months
  The primary objective of this study is to measure wide range of IOP values with the new tonometer and three comparator devices. The IOP value's unit of measure will be mmHg.

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - Vid d.o.o., Kromberk, Nova Gorica
  - Optika Mesec d.o.o., Bled, Občina Bled

IPD SHARING:
Plan to Share IPD: No